CLINICAL TRIAL: NCT03643367
Title: Sevoflurane Sedation: A Potentially Promising Immunomodulation in Patients With Septic Shock
Brief Title: Sevoflurane Sedation in Patients With Septic Shock
Acronym: SSiS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Münsterlingen (Other); Triemli Hospital (Other); Waid City Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSiS
Record Dates: First submitted 2017-06-20; First posted 2018-08-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Shock, Septic
Keywords: Sepsis; Septic Shock; Sevoflurane Conditioning
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Sevoflurane; Control Groups; Propofol

STUDY DESIGN:
Intervention Model Description: Patients with septic shock are intubated and ventilated and therefore need sedation. So far, most ICU centers use intravenously applied sedatives in these patients. In the proposed study, we will switch sedation from an intravenous to a volatile anesthetic for a short period of time (4 hours) to explore if sepsis markers improve within the following 120 hours upon sevoflurane conditioning.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be informed about their group assignments, technicians, processing the samples, will not have any access to ICU or patient charts (= double blind trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane Sedation (Experimental): Patients randomized into experimental group will be treated with sevoflurane during 4 hours
  Interventions: Drug: Sevoflurane
- Propofol Sedation (Active Comparator): Patients randomized into Control Group will get continued intravenous sedation with propofol
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Sevoflurane — Included patients, randomized in experimental group, intravenous sedation will be interrupted and followed by a 4 hour sedation with the volatile anesthetic sevoflurane.
  Arms: Sevoflurane Sedation
Drug: Control Group — Included patients randomized in control group, intravenouse sedation is continued with propofol
  Other Names: Propofol
  Arms: Propofol Sedation

SUMMARY:
Recent in vivo studies from others as well as the investigators group demonstrated that volatile anesthetics immunomodulate sepsis and improve outcome. Also, several clinical trials have convincingly shown that application of a volatile anesthetic provides protection in patients undergoing major surgery.

Patients with sepsis are intubated and ventilated and therefore need sedation. So far, most ICU centers use intravenously applied sedatives in these patients. In the proposed study, we will switch sedation from an intravenous to a volatile anesthetic for a short period of time to explore if sepsis markers improve within the following 120 hours upon sevoflurane conditioning.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will be conducted over a period of 48 months, to investigate if volatile anesthetics have a positive effect on the prognostic sepsis marker IL-6. All patients with septic shock are intubated, ventilated and sedated with an intravenous anesthetic. In this study, eligible patients diagnosed with septic shock will be randomized 1:1 to the 'volatile group' with interruption of the propofol infusion, followed by a 4-hour sedation with the volatile anesthetic sevoflurane, or a continuous intravenous sedation ('intravenous' =control group). In both groups, 'intravenous' and 'volatile', the inflammatory markers as well as clinical parameters will be determined. The investigators will explore if there is a difference between the course of sepsis markers of the two groups within 5 days after intervention in favor of the volatile group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18 to 80 years
* Intensive care Unit (ICU) patients with septic shock (despite fluid resuscitation vasopressors needed to maintain mean arterial pressure ≥65 millimeter of mercury (mmHg), and serum lactate >2mmol/l even with fluid application)
* Treatment of septic shock on ICU with vasopressors not longer than 12 hours
* Sedation and mechanical ventilation on ICU
* Female patients of childbearing potential with negative pregnancy test
* Informed Consent as documented by signature

Exclusion Criteria:

* Previous surgery and/or anesthesia (within last 7 days)
* Application of nitric oxide (NO)
* Suspected or known intolerance by history to volatile anesthetics (malignant hyperthermia)
* Immunosuppressive agents
* Systemic corticosteroids in the phase before hospitalization (> 10mg/d prednisone)
* Significant concomitant disease (acute cerebral vascular event, acute coronary syndrome, decompensated heart failure, acute pulmonary edema, major cardiac arrhythmia, seizure, burn, chronic kidney disease, end stage liver failure, neuromuscular disease)
* AIDS
* Autoimmune disease
* Organ transplant
* Subject with active malignancy receiving
* chemotherapy or radiation treatment within last 60 days
* Hepatitis B/C virus infection
* Anti-tumor necrosis factor (TNF) therapy
* Pregnancy and/or Breast feeding
* Use of cytokine absorber
* Enrollment in any other clinical trial during the course of this trial, 30 days prior to its beginning or 30 days after its completion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Concentration of interleukin-6 over time | 5 days
  To see if the interleukin-6 decreases under the influence of sevoflurane

SECONDARY OUTCOMES:
Pro-/anti-inflammatory mediators | 5 days
  effect on inflammatory/anti- inflammatory mediators
Vasopressor support | 5 days
  Use of vasopressor support (norepinephrine, dobutamine, vasopressin) will be determined.
Sequential organ failure score (SOFA Score) | 5 days
  Sepsis related organ failure score
Richmond Agitation Sedation Scale | 5 days
  A scale to measure the agitation or sedation level of a patient
Duration of mechanical ventilation | 28 days
  Time of mechanical ventilation
Mortality | 28 days
  Mortality information in intensive care unit and on the ward

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schlaepfer, PD, Principal Investigator — University of Zurich
Locations (4):
- Switzerland (4):
  - Kantonasspital Münsterlingen, Münsterlingen
  - Stadtspital Triemli, Zurich
  - University Hospital of Zurich, Zurich
  - Waidspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang BM, McLean AS, Dawes IW, Huang SJ, Lin RC. The use of gene-expression profiling to identify candidate genes in human sepsis. Am J Respir Crit Care Med. 2007 Oct 1;176(7):676-84. doi: 10.1164/rccm.200612-1819OC. Epub 2007 Jun 15. PMID 17575094
- [Background] Lu Y, Wang J, Yan J, Yang Y, Sun Y, Huang Y, Hu R, Zhang Y, Jiang H. Sevoflurane attenuate hypoxia-induced VEGF level in tongue squamous cell carcinoma cell by upregulating the DNA methylation states of the promoter region. Biomed Pharmacother. 2015 Apr;71:139-45. doi: 10.1016/j.biopha.2015.02.032. Epub 2015 Mar 3. PMID 25960229
- [Background] Klag T, Cantara G, Sechtem U, Athanasiadis A. Interleukin-6 Kinetics can be Useful for Early Treatment Monitoring of Severe Bacterial Sepsis and Septic Shock. Infect Dis Rep. 2016 Mar 21;8(1):6213. doi: 10.4081/idr.2016.6213. eCollection 2016 Mar 21. PMID 27103972
- [Background] Rios-Toro JJ, Marquez-Coello M, Garcia-Alvarez JM, Martin-Aspas A, Rivera-Fernandez R, Saez de Benito A, Giron-Gonzalez JA. Soluble membrane receptors, interleukin 6, procalcitonin and C reactive protein as prognostic markers in patients with severe sepsis and septic shock. PLoS One. 2017 Apr 5;12(4):e0175254. doi: 10.1371/journal.pone.0175254. eCollection 2017. PMID 28380034
- [Background] Tschaikowsky K, Hedwig-Geissing M, Braun GG, Radespiel-Troeger M. Predictive value of procalcitonin, interleukin-6, and C-reactive protein for survival in postoperative patients with severe sepsis. J Crit Care. 2011 Feb;26(1):54-64. doi: 10.1016/j.jcrc.2010.04.011. Epub 2010 Jun 19. PMID 20646905
- [Background] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Background] Kellner P, Muller M, Piegeler T, Eugster P, Booy C, Schlapfer M, Beck-Schimmer B. Sevoflurane Abolishes Oxygenation Impairment in a Long-Term Rat Model of Acute Lung Injury. Anesth Analg. 2017 Jan;124(1):194-203. doi: 10.1213/ANE.0000000000001530. PMID 27782948